CLINICAL TRIAL: NCT01915953
Title: A Clinical Evaluation of the OrSense Non-invasive Blood Hb/Hct Measurement Instrument, the Hemo-Monitor NBM200/MP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OrSense, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QD04.5.1-15
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-07

CONDITIONS: Anemia
Keywords: Accurte Hb noninvasive measurement
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- anemia: Measuring Hb valuse on anemia patients

SUMMARY:
The purpose of the study is to define the precision, accuracy and variability of the NBM-200 system in non invasive blood Hemoglobin (Hb) measurements relative to the laboratory blood analyzer by comparing two consecutive Hb values obtained by the NBM system to venous values.

DETAILED DESCRIPTION:
Each subject will be placed in a comfortable position in a temperature regulated room. Participants will have two consecutive non invasive (NBM) measurements taken which involves inserting the thumb into a ring shaped sensor. After each non invasive measurement the sensor will be removed. Each measurement takes approximately 85 seconds and involves the finger cuff inflating (to over systolic pressure) and deflating several times in quick successions in order to measure and calculate the Hb values. The two non invasive measurements will be performed using the same finger. After the NBM system testing is complete and recorded, the subject will have a venous (venipuncture) blood sample collected in order to provide two blood tests performed on two different models of routine automated complete blood count or Hb blood analyzers.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years and over

Exclusion Criteria:

* Participants under the age of 18 years
* Patients with significant deformity, degenerative changes or oedema of the fingers or hand
* Patients with localized infection, ulceration or skin breaks involving the fingers
* Patients with vascular disease or Raynaud's phenomenon affecting the fingers (vasospasm)
* Participants who are unable to give informed written consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematology pateints
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
compre the Hb values from the NBM200 series gainst the Hb from the lab blood analyser on Hematology pateints | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Korenberg, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Beer Yaacov, Israel, Israel